CLINICAL TRIAL: NCT00729807
Title: Treatment of Melanoma With Wild-type p53 and Detectable S100B Using Pentamidine: a Phase II Trial With Correlative Biomarker Endpoints
Brief Title: 0794GCC: Pentamidine in Treating Patients With Relapsed or Refractory Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed at the suggestion of DSMB prior to obtaining target enrollment
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-29873;HP-00040559; CDR0000602047 (Registry Identifier: PDQ (Physician Data Query)); HP-00047658 (Other: University of Maryland Human Research Protections Office); CINJ-090803 (Other: Cancer Institute of New Jersey); 0220090161 (Other: UMDNJ IRB Number); R21CA135624 (NIH)
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-06

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Pentamidine

STUDY DESIGN:
Intervention Model Description: This is an open label Phase II trial that will utilize a Simon two stage acquisition of patients with evaluable relapsed and/or refractory melanoma.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pentamidine (Experimental)
  Interventions: Drug: pentamidine

INTERVENTIONS:
Drug: pentamidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pentamidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well pentamidine works in treating patients with relapsed or refractory melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate in patients with relapsed or refractory melanoma that expresses wild-type p53 and S100 calcium binding protein B (S100B) treated with pentamidine.

Secondary

* To observe the effect of this drug on the expression of S100B and p21 in tumor biopsy samples.
* To observe the effect of this drug on S100B detectable in serum.
* To observe the time to progression in these patients.
* To assess the toxicities associated with the administration of this drug in these patients.

OUTLINE: Patients receive pentamidine IV over 2 hours 5 days a week for 2 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection periodically for correlative laboratory studies. Samples are assessed for p53 status and S100B, p53, and p21 expression by immunohistochemistry, polymerase chain reaction, western blotting, luminescence assay, and ELISA.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Relapsed or refractory disease
* Tumor expresses wild-type p53
* Measurable S100B by immunohistochemistry
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan
* Tumor amenable to biopsy
* Must have been evaluated for potentially curative resection
* No unstable or symptomatic brain metastases (e.g., seizures, headache related to tumor, or presence of neurologic deficits attributable to tumor)

  * Patients with stable brain metastases (by CT scan or MRI) are eligible provided they were treated with local therapy > 4 weeks ago AND do not require maintenance steroid treatment

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy > 12 weeks
* White Blood Cell count (WBC) ≥ 3,000/mcL
* Absolute Neutrophil Count (ANC) ≥ 1,500/mcL
* Platelet count ≥ 80,000/mcL
* Hemoglobin ≥ 8 g/dL
* Total bilirubin ≤ 1.5 times normal
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 times normal or creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* Able to take oral medications on a regular basis
* No history of allergic reactions attributed to pentamidine
* Mean Corrected QT Interval (QTc) ≤ 470 msec (with Bazett's correction) on screening ECG
* No history of familial long QT syndrome
* Proteinuria ≤ 1 on two consecutive dipsticks taken ≥ 1 week apart
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Hypertension
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Renal failure
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* Any number of prior chemotherapy regimens allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior radiotherapy or major surgery
* More than 30 days since prior participation in an investigational trial
* No concurrent medication that may markedly affect renal function (e.g., vancomycin, amphotericin, zoledronic acid)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Sausville, MD, PhD, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-treatment Evaluation: Following informed consent, patients will be scheduled for a biopsy of accessible tumor. The specimen will be assessed for p53 status by sequencing and S100B, p53, and p21 expression
Groups:
- Treatment Arm: Pentamidine isethionate will be administered at a dose of 4 mg/kg/day over 120 minutes each day, Monday - Friday for two weeks followed by a drug free period of 2 weeks.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Patients will receive 4 mg/kg/day IV pentamidine isethionate infused slowly over 2 hours on each treatment day. Each treatment cycle will consist of 2 weeks of therapy, five days per week, followed by 2 weeks of observation.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 63 [43 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate in Patients Treated With Pentamidine
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease, taking as reference the smallest sum of the longest diameter since the treatment started. (Therasse, P., Arbuck, S.G., Eisenhauer, E.A., Wanders, J., Kaplan, R.S., Rubinstein, J., Van Glabbeke, M., van Oosterom, A.T., Christian, M.C., Gwyther, S.G. (2000) J Natl Cancer Inst 92, 205-16)
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
Population: Six participants analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Pentamidine: Pentamidine isethionate will be administered at a dose of 4 mg/kg/day over 120 minutes each day, Monday - Friday for two weeks followed by a drug free period of 2 weeks.
Arm/Group | Pentamidine
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Number of Participants With Both p21 and S100B Expression in Accessible Tumor Biopsies Pre Pentamidine Exposure in Cycle 1
Description: Core Needle Tumor Biopsy
Time Frame: Pre-Study, an average of 12 days
Population: Only data for 1 site was analyzed for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Pentamidine
Number analyzed (Participants) | 4
Participants | 3

3. Secondary Outcome: Number of Participants With p21 and S100B Expression in Accessible Tumor Biopsies Post Pentamidine Exposure
Description: Core needle tumor biopsy - at Day 12 at first cycle of treatment
Time Frame: Day 12 Cycle 1
Population: Only 1 participant from 1 site had a biopsy collected and analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Pentamidine
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Expression of S100B Pre Pentamidine Exposure
Description: Serum for S100B
Time Frame: Pre-Study
Population: Only data for 1 site was analyzed for this outcome measure.
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Pentamidine
Number analyzed (Participants) | 4
pg/ml | 332.5 [116.5 to 5090]

5. Secondary Outcome: Expression of S100B
Description: Serum for S100B level
Time Frame: Cycle 1 Day 8, Cycle 1 Day 12, Cycle 2 Day 8, Cycle 2 Day 12
Population: Only data from 1 site was analyzed for this outcome measure
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Pentamidine
Number analyzed (Participants) | 4
pg/ml
  C1D8 | 450 [88.1 to 5679]
  C1D12 | 137 [74 to 5409]
  C2D8: number analyzed (Participants) | 2
  C2D8 | 142.1 [125 to 159.2]
  C2D12: number analyzed (Participants) | 1
  C2D12 | 150 [150 to 150]

6. Secondary Outcome: Number of Participants With Serious and Non Serious Adverse Events
Description: Metabolic Panel, Physical Exam, Vitals
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pentamidine
Number analyzed (Participants) | 6
Participants | 6

7. Secondary Outcome: Time to Progression
Description: Radiologic intervention using RECIST (x-ray, CT, MRI)
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: Every 8 weeks, assesed up to 6 months
Population: Only data for 1 site was analyzed for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Pentamidine
Number analyzed (Participants) | 3
days | 36 [36 to 51]

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=6)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) — Patient required hospitalization. Patient taken off treatment.
Infection (Infections and infestations) | 1 (1) — Patient required hospitalization. Patient's treatment was interrupted.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=6)
Anorexia (Gastrointestinal disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Blood in urine (Renal and urinary disorders) | 2 (2)
Creatinine (Renal and urinary disorders) | 2 (4)
Deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dry heaves (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Edema (Blood and lymphatic system disorders) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Fatigue (General disorders) | 3 (3)
Headache (General disorders) | 1 (1)
Heart palpitation (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (8)
Hypoalbuminemia (General disorders) | 1 (1)
Hypokalemia (General disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (6)
Hypotension (General disorders) | 2 (3)
Increase in GERD symptoms (Gastrointestinal disorders) | 1 (1)
Infiltration (General disorders) | 1 (2)
Insomnia (General disorders) | 1 (1)
Intermittent hypotension (Vascular disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Metallic taste in mouth (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Numbness of the face (Nervous system disorders) | 1 (2)
Proteinuria (General disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Reduced hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Upper back pain (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weakness (General disorders) | 2 (2)
Wound re-open (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Unable to reach the target number of participants needed before study was closed at the suggestion of DSMB

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No